CLINICAL TRIAL: NCT00010023
Title: A Phase I Study of Oral Fluoropyrimidine Capecitabine (Xeloda Roche) Combined With Intravenous Cisplatin in Patients With Advanced Cancer of the Digestive System
Brief Title: Capecitabine Combined With Cisplatin in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068434; P30CA016087 (NIH); NYU-9955; ROCHE-NYU-9955; NCI-G00-1908
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent non-small cell lung cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; small intestine adenocarcinoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; pulmonary carcinoid tumor; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; newly diagnosed carcinoma of unknown primary; carcinoma of the appendix; recurrent carcinoma of unknown primary; gastrointestinal stromal tumor; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Esophageal Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular; Gallbladder Neoplasms; Bile Duct Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Appendiceal Neoplasms; Neoplasms, Unknown Primary; Gastrointestinal Stromal Tumors; Salivary Gland Neoplasms | interventions — Capecitabine; Cisplatin

INTERVENTIONS:
Drug: capecitabine
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of capecitabine combined with cisplatin in treating patients who have locally advanced or metastatic solid tumors .

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity, maximum tolerated dose, and the recommended phase II dose of capecitabine and cisplatin in patients with locally advanced or metastatic cancer of the upper gastrointestinal tract (GI), head and neck, lung, breast, or carcinoma of unknown primary.
* Determine the toxic effects of this regimen in these patients.
* Evaluate possible antitumor effectiveness of this regimen in these patients.
* Determine the toxic effects of cisplatin and capecitabine at the recommended phase II dose in patients with cancer of the upper GI tract.
* Determine the overall survival, time to progression, and duration of response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of capecitabine.

Patients receive oral capecitabine twice daily for 5, 10, or 14 days. Patients also receive cisplatin IV on day 1 of each course. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). The recommended phase II dose is defined as the dose preceding the MTD, provided no more than 3 of 12 patients experience DLT at that dose. Twenty additional patients with cancer of the upper gastrointestinal tract receive treatment with cisplatin and capecitabine at the recommended phase II dose for at least 6 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 6 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 20-50 patients will be accrued for this study within 1-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or locally advanced inoperable carcinoma of the upper gastrointestinal tract, head and neck, lung, breast, or carcinoma of unknown primary
* Previously treated and/or resected primary tumors allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2 mg/dL*
* AST less than 3 times upper limit of normal (ULN)*
* Alkaline phosphatase no greater than 3 times ULN* NOTE: * Unless related to tumor (e.g., cholangiocarcinoma or hepatic metastases)

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* BUN no greater than 30 mg/dL* NOTE: * Unless related to tumor (e.g., cholangiocarcinoma or hepatic metastases)

Other:

* No other medical condition that could interfere with oral medication absorption
* No prior or concurrent malignancy except surgically cured carcinoma of the cervix or basal cell or squamous cell carcinoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 months since prior fluorouracil or cisplatin
* At least 3 weeks since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU Cancer Institute at New York University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Chen TT, Ryan T, Potmesil M, et al.: Cisplatin/capecitabine: tolerance and activity in patients with upper gastrointestinal cancers. [Abstract] American Society of Clinical Oncology 2004 Gastrointestinal Cancers Symposium, 22-24 January 2004, San Francisco, CA. A-53, 2004.